CLINICAL TRIAL: NCT02505568
Title: An Interventional, Open-label, Single Arm, Multicenter Study to Evaluate Efficacy and Safety of Infliximab in Subject With Moderate-to-Severe Refractory Intestinal Behcet's Disease
Brief Title: A Study to Evaluate Efficacy and Safety of Infliximab in Participant With Moderate-to-Severe Refractory Intestinal Behcet's Disease
Acronym: BEGIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR107121; REMICADEBEC3001 (Other: Janssen Korea, Ltd)
Record Dates: First submitted 2015-06-29; First posted 2015-07-22 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Behcet Disease
Keywords: Behcet Disease; Infliximab; Adult participants
MeSH Terms: conditions — Behcet Syndrome | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infliximab (Experimental): Participants will receive infliximab 5 milligram per kilogram (mg/kg) infusion at Week 0, Week 2, and Week 6 and will be evaluated for the induction phase at Week 8. Participants who complete the induction phase will continuously receive 5 mg/kg infliximab infusion at Week 14, Week 22, and Week 30 in the maintenance phase and will be evaluated at Week 32.
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Participants will receive infliximab 5 milligram per kilogram (mg/kg) infusion at Week 0, Week 2, and Week 6 for the induction phase. Participants who complete the induction phase will continuously receive 5 mg/kg infliximab infusion every 8 weeks up to week 32 in the maintenance phase.

SUMMARY:
The purpose of this study is to evaluate the efficacy of infliximab in induction regimen by assessing the mean decrease in Disease Activity Index for intestinal Behcet's disease (DAIBD) score of 20 or more in participants with active intestinal Behcet's disease who are refractory to conventional therapies.

DETAILED DESCRIPTION:
This is an open-label (all participants know the identity of the intervention), single arm, multicenter (when more than one hospital or medical school team work on a medical research study) study of Infliximab in participant with Moderate-to-Severe Refractory Intestinal Behcet's Disease. The study consists of 3 Phases: Screening Phase (4 weeks), induction Phase for 8 weeks, and maintenance Phase for 24 weeks extending from Week 0 (baseline), and a safety Follow up visit (Week 36 or approximately 6 weeks after the last administration of study drug). The duration of participation in the study for each participant is approximately 40 weeks. The mean decrease in Disease Activity Index for intestinal Behcet's disease (DAIBD) score of 20 or more will be evaluated primarily. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant had diagnosed of definite or probable intestinal Behcet's Disease (BD) prior to Screening
* Participant must have active intestinal BD, defined as; a) A baseline Disease Activity Index for intestinal Behcet's disease (DAIBD) score of greater than or equal to (>=) 40; b) Endoscopy with evidence of active intestinal BD (defined as ulcerations in the ileum and/or colon). The endoscopy must have occurred within 3 months prior to baseline
* Must either be currently receiving treatment with, or have a history of having failed to respond to, or tolerate, at least 1 of the following therapies as assessed by treating physician: oral corticosteroids, 6-mercaptopurine (6-MP), azathioprine (AZA), or methotrexate (MTX). a) Have no response to oral corticosteroids within the preceding 18 months; b) Have no response to 6-MP, AZA or MTX within the preceding 5 years
* Prior to the baseline, the following conditions must be met: a) If receiving 6-MP, AZA, or MTX must have been receiving it for at least 12 weeks, and the dose must be stable for at least 4 weeks; b) If 6-MP, AZA, or MTX have been recently discontinued, they must have been stopped for at least 4 weeks; c) If receiving oral 5-aminosalicylate (5-ASA) compounds or oral corticosteroids, the dose must have been stable for at least 2 weeks; d) If oral 5-ASA compounds or oral corticosteroids have been recently discontinued, they must have been stopped for at least 2 weeks; e) If receiving cyclosporine, the dose must have been stable for at least 6 weeks; f) If cyclosporine have been recently discontinued, they must have been stopped for at least 6 weeks
* Participant must be medically stable on the basis of physical examination, medical history, vital signs and 12-lead electrocardiogram (ECG) performed at Screening. If there are abnormalities, they must be consistent with the underlying illness in the study population, or the participant may be included only if the investigator judge the abnormalities from normal to be not clinically significant or to be appropriate. This determination must be recorded in the participant's source documents by the investigator

Exclusion Criteria:

* Participant has complications of intestinal BD such as symptomatic strictures or stenoses, short gut syndrome, central nervous system or vascular manifestation, or any other manifestation that might be anticipated to require surgery, could preclude the use of the DAIBD to assess response to therapy, or would possibly confound the ability to assess the effect of treatment with infliximab
* Participant currently has or is suspected to have an abscess. Recent cutaneous and perianal abscesses are not exclusionary if drained and adequately treated at least 3 weeks prior to baseline, or 8 weeks prior to baseline for intra-abdominal abscesses, provided that there is no anticipated need for any further surgery. Participants with active fistulas may be included if there is no anticipation of a need for surgery and there are currently no abscesses identified
* Participant has had any kind of bowel resection within 6 months or any other intra-abdominal surgery within 3 months prior to baseline
* Participant has a draining (ie, functioning) stoma or ostomy
* Participant has received any of the following prescribed medications or therapies within the specified period: a) Intravenous (IV) corticosteroids within 3 weeks prior to baseline; b) Other oral immunomodulatory agents (eg, 6-thioguanine (6-TG), tacrolimus, sirolimus, or mycophenolate mofetil) within 6 weeks prior to baseline; c) Non-biologic experimental or investigational agents within 4 weeks or within 5 half-lives of agent prior to baseline, whichever is longer; d) Other immunomodulatory biologic agents within 12 weeks or within 5 half-lives of agent prior to baseline, whichever is longer; e) Treatment with apheresis (eg, Adacolumn apheresis) or total parenteral nutrition (TPN) as a treatment for intestinal BD within 3 weeks prior to baseline

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-07-22 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
The Mean Decrease in Disease Activity Index for Intestinal Behcet's Disease (DAIBD) Score of 20 or More From Baseline at Week 8 | Baseline and Week 8
  The DAIBD will be assessed by collecting information on 8 different intestinal BD-related variables. These 8 variables are: fever, abdominal mass, abdominal tenderness, intestinal complications, extraintestinal manifestations, general well-being, abdominal pain, and total number of liquid stools. The last 3 variables are scored over 7 days by the participant on a diary card. Abdominal pain will be measured using the 11-point numeric rating scale (NRS) to standardize the evaluation of pain and the result of 11-point NRS will be divided into 4 grades (none, mild, moderate, severe) to fill out the DAIBD. where, None indicate 0; Mild indicate 1-3; Moderate indicate 4-6; Severe indicate 7-10.

SECONDARY OUTCOMES:
Percentage of Participant With Clinical Response by Disease Activity Index for Intestinal Behcet's Disease (DAIBD) at Week 8 and 32 | At Week 8 and 32
  The DAIBD will be assessed by collecting information on 8 different intestinal BD-related variables. These 8 variables are: fever, abdominal mass, abdominal tenderness, intestinal complications, extraintestinal manifestations, general well-being, abdominal pain, and total number of liquid stools. The last 3 variables are scored over 7 days by the participant on a diary card. Abdominal pain will be measured using the 11-point numeric rating scale (NRS) to standardize the evaluation of pain and the result of 11-point NRS will be divided into 4 grades (none, mild, moderate, severe) to fill out the DAIBD. where, None indicate 0; Mild indicate 1-3; Moderate indicate 4-6; Severe indicate 7-10.
Percentage of Participant With Crohn's Disease Activity Index (CDAI) 70 Response at Week 8 and 32 | At Week 8 and 32
  The CDAI will be assessed by collecting information on 8 different Crohn's disease-related variables. These 8 variables are: extraintestinal manifestations, abdominal mass, weight, hematocrit, use of antidiarrheal drug(s) and/or opiates, total number of liquid stools, abdominal pain/cramping, and general well-being. The last 3 variables are scored over 7 days by the participant on a diary card. The CDAI 70-response is defined as a reduction from baseline in the CDAI score of greater than or equal to (>=) 70 points.
Change in Crohn's Disease Activity Index (CDAI) Score From Baseline at Week 8 and 32 | Baseline, Week 8 and 32
  The CDAI will be assessed by collecting information on 8 different Crohn's disease-related variables. These 8 variables are: extraintestinal manifestations, abdominal mass, weight, hematocrit, use of antidiarrheal drug(s) and/or opiates, total number of liquid stools, abdominal pain/cramping, and general well-being. The last 3 variables are scored over 7 days by the participant on a diary card.
Change in C -Reactive Protein (CRP) Concentration From Baseline at Week 8 and 32 | Baseline, Week 8 and 32
  The CRP has been demonstrated to be useful as a marker of inflammation in patients with inflammatory bowel disease (IBD). In Behcet's Disease (BD), CRP concentrations in active disease participants have been found to be higher than those in inactive participants. Blood samples for the measurement of CRP will be collected from all participants. CRP will be assayed using a validated, high sensitivity CRP assay.
Change in Disease Activity Index for Intestinal Behcet's Disease (DAIBD) Score From Baseline at Week 32 | Baseline and Week 32
  The DAIBD will be assessed by collecting information on 8 different intestinal BD-related variables. These 8 variables are: fever, abdominal mass, abdominal tenderness, intestinal complications, extraintestinal manifestations, general well-being, abdominal pain, and total number of liquid stools. The last 3 variables are scored over 7 days by the participant on a diary card. Abdominal pain will be measured using the 11-point numeric rating scale (NRS) to standardize the evaluation of pain and the result of 11-point NRS will be divided into 4 grades (none, mild, moderate, severe) to fill out the DAIBD. where, None indicate 0; Mild indicate 1-3; Moderate indicate 4-6; Severe indicate 7-10.
Percentage of Participant With Clinical Remission (Disease Activity Index for Intestinal Behcet's Disease [DAIBD] Score less than or equal to [<=] 19) at Week 32 | Week 32
  The DAIBD will be assessed by collecting information on 8 different intestinal BD-related variables. These 8 variables are: fever, abdominal mass, abdominal tenderness, intestinal complications, extraintestinal manifestations, general well-being, abdominal pain, and total number of liquid stools. The last 3 variables are scored over 7 days by the participant on a diary card. Abdominal pain will be measured using the 11-point numeric rating scale (NRS) to standardize the evaluation of pain and the result of 11-point NRS will be divided into 4 grades (none, mild, moderate, severe) to fill out the DAIBD. where, None indicate 0; Mild indicate 1-3; Moderate indicate 4-6; Severe indicate 7-10.
Period Needed to Reach Clinical Remission From Baseline at Week 32 | Up to Week 32
  The duration for participants required to reach clinical remission will be analysed.
Percentage of Participants With Mucosal Healing at Week 32 | Week 32
  Mucosal healing will be assessed using endoscopy (ileocolonoscopy) in consenting participants. A video ileocolonoscopic examination will be performed according to the study reference manual provided to each site, at Screening and Week 32. Investigators will measure the longest diameter (none, >= 1 centimeter [cm] to less than [<] 2 cm, >= 2 cm to < 3, >= 3 cm) of ileum and/or colon largest open ulcer and assess mucosal healing in 4 grades compared to the baseline according to the following; Grade 0: Mucosal healing; Grade 1: marked improvement (reduction to <= 1/4); Grade 2: improvement (reduction to <= 1/2 - > 1/4); Grade 3: no change or worse (reduction less than 1/2 or expansion).
Number of Participants with Adverse Events (AEs) and Serious AEs | Up to Week 36
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd Clinical Trial, Study Director — Janssen Korea, Ltd
Locations (5):
- South Korea (5):
  - Busan
  - Daegu
  - Gangwon-do
  - Gyeonggi-do
  - Seoul

REFERENCES:
- [Derived] Cheon JH, Kim HS, Han DS, Kim SK, Shin SJ, Kim JS, Ye BD, Song GA, Lee Y, Kim Y, Lee Y, Kim WH; BEGIN Study Group. Efficacy and Safety of Infliximab in Intestinal Behcet's Disease: A Multicenter, Phase 3 Study (BEGIN). Gut Liver. 2023 Sep 15;17(5):777-785. doi: 10.5009/gnl220278. Epub 2022 Dec 29. PMID 36578194
- See also: An Interventional, Open-label, Single Arm, Multicenter Study to Evaluate Efficacy and Safety of Infliximab in Subjects with Moderate-to-Severe Refractory Intestinal Behcet's Disease — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR107121&attachmentIdentifier=dda5b9ac-dbb4-49d2-8544-5f820fd729e3&fileName=CR107121_CSR.pdf&versionIdentifier=